CLINICAL TRIAL: NCT03841851
Title: Aesthetic Outcome of Immediate Implant Placement With Immediate Loading With and Without Sub Epithelial Connective Tissue Graft
Brief Title: Immediate Implant Placement With Immediate Loading With and Without Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Habib, principle investigator(doctor), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: cairo univ
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pateint With Badely Decayed Anterior Teeth

STUDY DESIGN:
Intervention Model Description: This study will be conducted on patients with badely decayed teeth in aesthetic zone and need immediate fixed restoration .
  This study is to be conducted in Dental Implant Clinic, Faculty of Dentistry, Cairo University, Egypt.
  All the patients will be entailed about the study and given their approval to participate on written consent.
Who Masked: Participant, Investigator
Masking Description: Each patient will be given acode by the researcher and the observers will be blind to which group this case belong
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- temporization without soft tissue graft (No Intervention): * Local anesthesia will be injected intra-orally at the implant site.
  * Atraumatic extraction of badley decayed teeth in the aesthetic area
  * traditional drilling for immediate implant placement .
  * immediate temporization .
- temporization with soft tissue graft (Active Comparator): * Local anesthesia will be injected intra-orally at the implant site.
  * Atraumatic extraction of badley decayed teeth in the aesthetic area
  * traditional drilling for immediate implant placement .
  * immediate temporization .
  * subepithelial connective tissue graft from the palate .
  Interventions: Procedure: sub epithelial connective tissue graft

INTERVENTIONS:
Procedure: sub epithelial connective tissue graft — * Local anesthesia will be injected intra-orally at the implant site.
  * Atraumatic extraction of badley decayed teeth in the aesthetic area traditional drilling for immediate implant placement .
  * immediate temporization .
  * subepithelial connective tissue graft from the palate
  Arms: temporization with soft tissue graft

SUMMARY:
extraction of badely decayed anterior teeth immediate implant placement with immediate temporaization

DETAILED DESCRIPTION:
Intra-operative procedure:

Local anesthesia will be injected intra-orally at the implant site. Atraumatic extraction of badley decayed teeth in the aesthetic area .

For group A :

traditional drilling for immediate implant placement . immediate temporization .

For group B :

traditional drilling for immediate implant placement . immediate temporization . subepithelial connective tissue graft from the palate .

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable maxillary anterior teeth indicated for implant placement.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Patients with systemic disease that may affect bone quality.
* Patients with poor oral hygiene and active periodontal diseases.
* Heavy smokers more than 20 cigarettes per day.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Pink esthetics | every 2 weeks for 3 months
  evaluation of esthetic outcome using pink esthetic score

IPD SHARING:
Plan to Share IPD: No
Local anesthesia will be injected intra-orally at the implant site. Atraumatic extraction of badley decayed teeth in the aesthetic area .
  For group A :
  * traditional drilling for immediate implant placement .
  * immediate temporization .
  For group B :
  * traditional drilling for immediate implant placement .
  * immediate temporization .
  * subepithelial connective tissue graft from the palate

REFERENCES:
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184
- [Background] Salama H, Salama MA, Li TF, Garber DA, Adar P. Treatment planning 2000: an esthetically oriented revision of the original implant protocol. J Esthet Dent. 1997;9(2):55-67. doi: 10.1111/j.1708-8240.1997.tb00919.x. PMID 9468854
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Adell R, Eriksson B, Lekholm U, Branemark PI, Jemt T. Long-term follow-up study of osseointegrated implants in the treatment of totally edentulous jaws. Int J Oral Maxillofac Implants. 1990 Winter;5(4):347-59. PMID 2094653
- [Background] Schnitman PA, Wohrle PS, Rubenstein JE, DaSilva JD, Wang NH. Ten-year results for Branemark implants immediately loaded with fixed prostheses at implant placement. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):495-503. PMID 9274078
- [Background] Testori T, Meltzer A, Del Fabbro M, Zuffetti F, Troiano M, Francetti L, Weinstein RL. Immediate occlusal loading of Osseotite implants in the lower edentulous jaw. A multicenter prospective study. Clin Oral Implants Res. 2004 Jun;15(3):278-84. doi: 10.1111/j.1600-0501.2004.01013.x. PMID 15142089
- [Background] Redemagni M, Cremonesi S, Garlini G, Maiorana C. Soft tissue stability with immediate implants and concave abutments. Eur J Esthet Dent. 2009 Winter;4(4):328-37. PMID 20111758
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Sanz M, Cecchinato D, Ferrus J, Pjetursson EB, Lang NP, Lindhe J. A prospective, randomized-controlled clinical trial to evaluate bone preservation using implants with different geometry placed into extraction sockets in the maxilla. Clin Oral Implants Res. 2010 Jan;21(1):13-21. doi: 10.1111/j.1600-0501.2009.01824.x. Epub 2009 Nov 18. PMID 19922492
- [Background] Cosyn J, Hooghe N, De Bruyn H. A systematic review on the frequency of advanced recession following single immediate implant treatment. J Clin Periodontol. 2012 Jun;39(6):582-9. doi: 10.1111/j.1600-051X.2012.01888.x. Epub 2012 Apr 18. PMID 22509794